CLINICAL TRIAL: NCT06182683
Title: Concurrent OPTIcal Coherence Tomography and frActional Flow REserve-guided Therapeutic Intervention in Patients With Coronary Artery Disease (OPTICARE-CAD)
Brief Title: Concurrent OCT and FFR-guided PCI in CAD
Acronym: OPTICARE-CAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Responsible Party: Principal Investigator, Kang Dong Oh, Assistant Professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPTICARE-CAD_v1
Record Dates: First submitted 2023-11-28; First posted 2023-12-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Coronary Artery Disease; Image; Atheroscleroses, Coronary
Keywords: Optical coherence tomography; Fractional flow reserve; Angiography; Coronary artery disease; Percutaneous coronary intervention; Drug-eluting stent
MeSH Terms: conditions — Coronary Artery Disease | interventions — Tomography, Optical Coherence; Coronary Angiography

STUDY DESIGN:
Intervention Model Description: Prospective, randomized open-label clinical trial
Masking Description: No blinding process, open label design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Angiography-guided PCI group (Active Comparator): This group of patients are intended to undergo PCI with conventional angiography-guidance. Procedural optimization determined by angiographic assessment.
  Interventions: Diagnostic Test: Coronary angiography
- Concurrent OCT/FFR-guided PCI group (Experimental): This group of patients are intended to undergo PCI with concurrent OCT/FFR-guidance. Procedural optimization determined by OCT and FFR assessment.
  Interventions: Diagnostic Test: optical coherence tomography and fractional flow reserve; Diagnostic Test: Coronary angiography

INTERVENTIONS:
Diagnostic Test: optical coherence tomography and fractional flow reserve — The assessment of pre-procedural lesions and optimization status of implanted stents will involve both intracoronary imaging and physiological indices.
  Arms: Concurrent OCT/FFR-guided PCI group
Diagnostic Test: Coronary angiography — The assessment of pre-procedural lesions and optimization status of implanted stents will be determined by conventional coronary angiography

SUMMARY:
The present study is a prospective randomized clinical trial aimed to compare the therapeutic strategy of angiography-guided versus concurrent OCT/FFR-guided intervention in patients with coronary artery disease.

DETAILED DESCRIPTION:
Most previous clinical trials have assessed various interventional strategies guided by intravascular imaging (intravascular imaging-guided PCI), fractional flow reserve (FFR-guided PCI), or conventional angiography (angiography-guided PCI) to compare differences in treatment outcomes. Until now, it remains unclear whether optimizing procedures based on both intravascular imaging and fractional flow reserve indices would lead to improved treatment outcomes compared to PCI guided solely by conventional angiography. Moreover, there are no studies comparing a treatment strategy that combines optical coherence tomography (OCT) and FFR to angiography-guided procedures. Hence, this study aims to compare the clinical effectiveness and therapeutic impact of concurrent guidance using FFR and OCT in patients undergoing coronary artery stent implantation, as compared to procedures guided solely by conventional angiography.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than 19 years old
2. Patients undergoing coronary stent implantation for stable angina or acute coronary syndrome
3. Patients provided on informed consent

Exclusion Criteria:

1. Individuals with a history of increased bleeding tendencies or hematologic disorders
2. Presented with refractory cardiogenic shock
3. Individuals with a history of stent thrombosis
4. Expected life expectancy of less than 1 year
5. Left ventricular ejection fraction (LVEF) ≥ 20%
6. Women who are breastfeeding, pregnant, or planning to become pregnant
7. Deemed unsuitable for participation by the investigator
8. Patients unwilling to participate in the clinical trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of target vessel failure (TVF) | 1-year
  a composite endpoint of cardiac death, target vessel-related non-fatal myocardial infarction, clinically driven-target vessel revascularization

SECONDARY OUTCOMES:
Rate of all-cause mortality | 1-year
  cardiac and non-cardiac death
Rate of any myocardial infarction (MI) | 1-year
  myocardial infarction due to target vessel and non-target vessel failure
Rate of clinically-driven target vessel revascularization (TVR) | 1-year
  clinically-driven target vessel revascularization
Rate of any revascularization | 1-year
  clinically-driven target lesion and non-target lesion revascularization
Rate of stent thrombosis (acute, subacute, late, very late) | 1-year
  stent thrombosis based on presenting time after the index procedure
Rate of BARC-defined bleeding | 1-year
  clinically-relevant bleeding event based on BARC classification

OTHER OUTCOMES:
FFR optimization rate | Immediately after index procedure
  1) Post-PCI FFR ≥ 0.90, or 2) Post-PCI FFR (LAD) ≥ 0.82, or 3) Post-PCI FFR (non-LAD) ≥ 0.88, 4) Stent-segment ΔFFR ≤0.05
OCT optimization rate | Immediately after index procedure
  1) Post-PCI MSA ≥ 4.5 mm2, and 2) Post-PCI expansion ≥ 80%

CONTACTS AND LOCATIONS:
Overall Officials: Dong Oh Kang, MD, PhD, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will be available to qualified researchers only upon reasonable request and appropriate proposal to the principal investigator.

REFERENCES:
- [Background] Johnson TW, Raber L, di Mario C, Bourantas C, Jia H, Mattesini A, Gonzalo N, de la Torre Hernandez JM, Prati F, Koskinas K, Joner M, Radu MD, Erlinge D, Regar E, Kunadian V, Maehara A, Byrne RA, Capodanno D, Akasaka T, Wijns W, Mintz GS, Guagliumi G. Clinical use of intracoronary imaging. Part 2: acute coronary syndromes, ambiguous coronary angiography findings, and guiding interventional decision-making: an expert consensus document of the European Association of Percutaneous Cardiovascular Interventions. Eur Heart J. 2019 Aug 14;40(31):2566-2584. doi: 10.1093/eurheartj/ehz332. PMID 31112213
- [Background] Lawton JS, Tamis-Holland JE, Bangalore S, Bates ER, Beckie TM, Bischoff JM, Bittl JA, Cohen MG, DiMaio JM, Don CW, Fremes SE, Gaudino MF, Goldberger ZD, Grant MC, Jaswal JB, Kurlansky PA, Mehran R, Metkus TS Jr, Nnacheta LC, Rao SV, Sellke FW, Sharma G, Yong CM, Zwischenberger BA. 2021 ACC/AHA/SCAI Guideline for Coronary Artery Revascularization: Executive Summary: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2022 Jan 18;145(3):e4-e17. doi: 10.1161/CIR.0000000000001039. Epub 2021 Dec 9. PMID 34882436
- [Background] Collison D, Didagelos M, Aetesam-Ur-Rahman M, Copt S, McDade R, McCartney P, Ford TJ, McClure J, Lindsay M, Shaukat A, Rocchiccioli P, Brogan R, Watkins S, McEntegart M, Good R, Robertson K, O'Boyle P, Davie A, Khan A, Hood S, Eteiba H, Berry C, Oldroyd KG. Post-stenting fractional flow reserve vs coronary angiography for optimization of percutaneous coronary intervention (TARGET-FFR). Eur Heart J. 2021 Dec 1;42(45):4656-4668. doi: 10.1093/eurheartj/ehab449. PMID 34279606